CLINICAL TRIAL: NCT06349642
Title: Observational Basket Trial to Collect Tissue to Develop and Train a Live Tumor Diagnostic Platform
Brief Title: Immune Checkpoint Inhibitor Response in Solid Tumors Using a Live Tumor Diagnostic Platform
Acronym: ELEPHAS-04
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Elephas Biosciences Corporation (Unknown)
Responsible Party: Sponsor
Other Study IDs: MC230901; NCI-2024-02979 (Registry Identifier: CTRP (Clinical Trials Reporting Program)); 23-008413 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Early Stage Triple-Negative Breast Carcinoma; Metastatic Bladder Urothelial Carcinoma; Metastatic Cervical Carcinoma; Metastatic Clear Cell Renal Cell Carcinoma; Metastatic Colorectal Carcinoma; Metastatic Endometrial Carcinoma; Metastatic Esophageal Carcinoma; Metastatic Liver Carcinoma; Metastatic Lung Non-Small Cell Carcinoma; Metastatic Malignant Skin Neoplasm; Metastatic Malignant Solid Neoplasm; Resectable Lung Non-Small Cell Carcinoma; Early Stage Lung Non-Small Cell Carcinoma; Resectable Malignant Solid Neoplasm; Resectable Triple-Negative Breast Carcinoma; Stage III Renal Cell Cancer AJCC v8; Stage IV Cervical Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8; Stage IV Uterine Corpus Carcinoma or Carcinosarcoma AJCC v8; Recurrent Cervical Carcinoma; Recurrent Colorectal Carcinoma; Recurrent Endometrial Carcinoma; Recurrent Esophageal Carcinoma; Recurrent Liver Carcinoma; Recurrent Lung Non-Small Cell Carcinoma; Recurrent Malignant Skin Neoplasm; Recurrent Malignant Solid Neoplasm
MeSH Terms: conditions — Uterine Cervical Neoplasms; Clear-cell metastatic renal cell carcinoma; Colorectal Neoplasms; Endometrial Neoplasms; Esophageal Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Non-Small-Cell Lung; Skin Neoplasms; Neoplasm Metastasis; Carcinoma, Renal Cell; Carcinosarcoma | interventions — Blood Specimen Collection; Specimen Handling; Tissue Banks

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens will only be retained for future research if participant grants permission. Research specimen collection kits for optional blood samples will be created and managed by the Mayo Clinic Biospecimen Accessioning and Processing lab. Research tissue samples will be collected at the time of the patient's standard of care biopsy, or if the standard of care biopsy has already occurred then a research only biopsy will be scheduled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients undergo tissue biopsy and may optionally undergo blood sample collection and have their medical records reviewed on study. Patients receive standard treatment with checkpoint inhibitors during the study and undergo standard tumor assessments during screening and follow-up.
  Interventions: Procedure: Biospecimen Collection; Procedure: Tissue Collection

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo optional research blood sample.
  Other Names: Blood Draw; Specimen Collection
Procedure: Tissue Collection — Tissue specimen collection will be completed with your scheduled standard of care biopsy if possible. If standard of care biopsy is already completed or the research biopsy wasn't collected at the time as your standard of care biopsy, then the research biopsy will be scheduled for a different day for research purposes only.

SUMMARY:
This study is being done to collect tissue samples to test how accurately a tumor response platform, Elephas, can predict clinical response across multiple types of immunotherapies, chemoimmunotherapy and tumor types.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet one of the following criteria:

* Subjects suspected of or diagnosed with the following Stage IV/metastatic or recurrent malignancies:

  * Lung: Non-small Cell Lung Cancer (NSCLC)
  * Skin: Cutaneous Malignancy, excluding Uveal Melanoma
  * Esophageal Cancer
  * Cervical Cancer
  * Endometrial Cancer
  * Colon Cancer: Mismatch repair deficient (dMMR) CRC only
  * All solid tumors with high tumor mutation burden (TMB)
  * All solid tumors that are microsatellite instability high (MSI-H)
  * All mismatch repair deficient (dMMR) solid tumors
  * Liver Cancer
  * Any solid tumor with measurable disease that is eligible for pure ICI therapy or that the clinician plans to treat with immune checkpoint inhibitor (ICI) therapy. NOTE: This can be in the setting of a trial, compassionate use, or the use of appropriate laboratory developed tests (LDTs) that, per clinician, render the patient eligible for ICI therapy, either frontline or a later line.

OR

* Subjects suspected of or diagnosed with the following Stage III per provider discretion or IV/metastatic malignancies:

  * Kidney: Clear Cell Renal Cell Carcinoma (ccRCC)
  * Bladder: Urothelial Carcinoma (UC)
  * Any solid tumor with measurable disease that is eligible for pure ICI therapy or that the clinician plans to treat with ICI therapy. NOTE: This can be in the setting of a trial, compassionate use, or the use of appropriate LDT tests that per clinician, render the patient eligible for ICI therapy, either frontline or a later line

OR

* Patients who will be receiving neoadjuvant CPI for the following resectable early-stage malignancies:

  * Breast Cancer: Triple negative breast cancer (TNBC)
  * Lung: Non-small cell lung cancer (NSCLC)

    * NOTE: Patients with suspected NSCLC who would be eligible for neoadjuvant checkpoint inhibitor (CPI) are eligible to enroll per provider discretion
  * Any solid tumor that is eligible for pure ICI therapy or that the clinician plans to treat with ICI therapy. NOTE: This can be in the setting of a trial, compassionate use, or the use of appropriate LDT tests that per clinician, render the patient eligible for ICI therapy, either frontline or a later line
* LOCALLY ADVANCED/METASTATIC PATIENTS: Measurable disease as defined per protocol NOTE: Tumor lesions in a previously irradiated area are not considered measurable disease; Disease that is measurable by physical examination only is not eligible.
* NEOADJUVANT PATIENTS: Subjects must be eligible based on investigator discretion to receive approved CPI therapy.
* Subjects who are newly diagnosed or have suspected cancer must be treatment-naïve at the time of biopsy.
* Subjects who are Stage I, II, or III and have progressed to metastatic cannot have received any anti-cancer treatment for at least 2 - 4 weeks (depending upon the washout period of prior anti-cancer treatment) prior to biopsy as per the agents used.
* ECOG Performance Status (PS) 0, 1 or 2.
* Negative pregnancy test done ≤7 days prior to enrollment, for persons of childbearing potential only
* Female subjects must not be pregnant or breastfeeding and must use appropriate methods of contraception when applicable.
* Subjects must be clinically able, at investigator discretion, and willing to undergo either:

  * additional biopsy passes during their standard of care biopsy, OR
  * a biopsy for research only, if applicable.
  * NOTE: These additional biopsies may either be collected from the primary tumor or a metastatic site amenable to biopsies per the clinician.
* Subjects with a known secondary cancer diagnosis are eligible to participate if participation does not interfere with systemic anti-cancer standard of care treatment for suspected primary diagnosis.
* Provide written informed consent

Exclusion Criteria:

* Pregnant women because this study involves a greater than minimal risk procedure (biopsy)
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety for the biopsy
* Immunocompromised patients and patients known to be HIV positive and currently receiving antiretroviral therapy

  * NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Uncontrolled intercurrent illness including, but not limited to:

  * ongoing or active infection
  * psychiatric illness/social situations that would limit compliance with study requirements
* Subjects who are enrolled or plan to be enrolled in a blinded cancer therapeutic treatment trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at Mayo Clinic in Rochester who are suspected of or diagnosed with Stage III or IV/metastatic cancer or receiving neoadjuvant (pre-operative) checkpoint inhibitors (CPI) for a resectable early stage of solid malignancies
Sampling Method: Non-Probability Sample
Enrollment: 324 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the Elephas Score for predicting clinical response in neoadjuvant patients | Up to 3 years
  Assessed based on pathologic complete response (pCR) during checkpoint inhibitor (CPI) treatment. Clinical non-response will be defined as non-pathological complete response. Patients who cannot have pathologic complete response determined will be excluded from the primary analysis.
Accuracy of the Elephas Score for predicting clinical response in locally advanced/metastatic patients | Up to 3 years
  Assessed based on Response Evaluation Criteria In Solid Tumors (RECIST) score for best overall response [complete response (CR) or partial response (PR)] during checkpoint inhibitor (CPI) treatment. Clinical non-response will be defined as either stable disease (SD) or disease progression (PD). Patients who cannot have best response determined will be excluded from the primary analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Dev Mukhopadhyay, PhD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Phoenix, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramasubramanian TS, Adstamongkonkul P, Scribano CM, Johnson C, Caenepeel S, Hrycyniak LCF, Vedder L, Dana N, Baltes C, Browning T, Chen YI, Dietz T, Flietner E, Kaplewski N, Kellner A, Korrer M, Liu C, Marhefke N, McDonnell P, Nasreen A, Pope V, Prasad A, Richardson J, Schneider S, Schultz M, Sood C, Sunil A, von Euw E, Wait E, Wargowski E, Advani P, Broome B, Bruckbauer A, Godwin A, Kokabi N, Martin R, Robaina M, Toia G, Routh J, Friedl A, Eliceiri K, Szulczewski M, Johnson S, Oliner J, Galon J, Capitini C, Mukhopadhyay D, Taube J, Braun D, Gierman HJ. A live tumor fragment platform to assess immunotherapy response in core needle biopsies while addressing challenges of tumor heterogeneity. bioRxiv [Preprint]. 2025 Jul 18:2025.07.18.663728. doi: 10.1101/2025.07.18.663728. PMID 40791544
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials